CLINICAL TRIAL: NCT02197091
Title: A Health Services Research Study to Evaluate Communication Effectiveness in Oncology Treatment
Brief Title: Communication Effectiveness in Cancer Treatment
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00028889; NCI-2014-01478 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB00028889; CCCWFU #99514 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2014-07-21; First posted 2014-07-22 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (communication in oncology treatment): Patients complete questionnaires, including the FACIT-TS-G, the FACIT-Sp12, the MOS-SSS, and the DT. Doctors also complete a questionnaire. Patients' medical records may be reviewed, if necessary.
  Interventions: Other: questionnaire administration; Other: medical chart review

INTERVENTIONS:
Other: questionnaire administration — Ancillary studies
Other: medical chart review — Ancillary studies
  Other Names: chart review

SUMMARY:
This pilot research trial studies communication effectiveness in cancer treatment. Studying how well patients and their doctors communicate about the treatment being given for cancer may help improve the decisions that patients and physicians make together.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of measuring discrepancies between patient and physician perceptions about the intent of therapy.

SECONDARY OBJECTIVES:

I. To explore possible correlation between various patient satisfaction indicators and discrepant patient perceptions about their care.

II. To gather exploratory data on patient characteristics that might correlate with discrepant patient perceptions about their care.

OUTLINE:

Patients complete questionnaires, including the Functional Assessment of Cancer Therapy-Treatment Satisfaction (FACIT-TS-G), the Functional Assessment of Cancer Therapy-Spiritual Well Being (FACIT-Sp12), the Medical Outcomes Study Social Support Survey (MOS-SSS), and the Distress Thermometer (DT). Doctors also complete a questionnaire. Patients' medical records may be reviewed, if necessary.

After completion of study, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of cancer
* Patients must have been in active therapy for cancer for at least one month or have a scheduled surgical treatment of their cancer
* Ability to understand and the willingness to sign an institutional review board (IRB)-approved informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults receiving cancer treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Patient perceptions about the nature of their therapy and diagnosis | Baseline
  The precision of agreement between patient's and doctor's responses about the intent of therapy will be assessed. The level of agreement between the questions as answered by the patient on the Prognosis Instrument and by the doctor on the Doctor Questionnaire will be assessed. Agreement will be measured as either "yes" (meaning the doctor and patient responses match exactly) or "no" (any other combination, if both doctor and patient responded). The primary measure of agreement will be the Kappa statistic; the Kappa and its corresponding 95% confidence interval (CI) will be reported.
Feasibility, as assessed by accrual rate | Up to 5 years
  Accrual will be estimated as the number of patients accrued divided by the months of accrual. A 95% confidence interval for the monthly accrual will be calculated based on the Poisson distribution.
Feasibility, as assessed by participation rate | Up to 5 years
  The participation rate will be estimated as the number of patients who are participants divided by the number eligible. This estimate will be calculated separately by cancer type to see what cancer types are more or less likely to participate. An exact 95% CI will be calculated for this estimate of each cancer type.

SECONDARY OUTCOMES:
Incidence of discrepancies between patient perceptions and the clinical record | Baseline
  The FACIT-TS-G, FACIT-Sp12, MOS-SSS, and DT instruments will be used to see if there might be a relationship between the observed scores and discrepancies in the answers provided by patients and the clinical record. Patient characteristics will be assessed for differences between the two records. Means, standard deviations, and medians will be calculated for each of the scores, stratified by discrepancy type for those who do not match and those who match perfectly. These data will be analyzed by analysis of variance.

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Duckworth, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States